CLINICAL TRIAL: NCT06208358
Title: Brain Mechanism of Disrupted Interpersonal Interaction in Gaming Disorder Affecting Cognitive Control and Its Hierarchical Multidimensional Evaluation Intervention
Brief Title: A Study for the Disrupted Interpersonal Interaction Among Gaming Disorder Individuals and Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NZhong-006
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Gaming Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Active Comparator): Device: Transcranial Alternating Current Stimulation In recent years, transcranial alternating current stimulation (tACS) has been widely used to regulate brain neural activity and improve cognitive function because of its non-invasive, portable, and easy-to-operate characteristics. tACS can effectively improve 9 cognitive functions, including visual attention, working memory, long-term memory, executive control, fluid intelligence, learning, decision-making, motor learning, and motor memory
  Interventions: Device: tACS
- sham tACS (Sham Comparator): Device: Transcranial Alternating Current Stimulation In recent years, transcranial alternating current stimulation (tACS) has been widely used to regulate brain neural activity and improve cognitive function because of its non-invasive, portable, and easy-to-operate characteristics. tACS can effectively improve 9 cognitive functions, including visual attention, working memory, long-term memory, executive control, fluid intelligence, learning, decision-making, motor learning, and motor memory
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — We aim to use tACS devices to improve the disrupted interpersonal interaction among gaming disorder individuals.

SUMMARY:
Aiming at the major problems of unclear brain mechanism of gaming disorder and lack of effective assessment intervention tools, this project started by exploring the brain mechanism of abnormal interpersonal interaction and cognitive control deficit promoting and accelerating the development of gaming disorder, adopted a prospective cohort study design, combined with multi-modal brain functional imaging, cognitive function, social psychological assessment, and other means. To clarify the brain mechanism and outcome of gaming disorder. Based on the preliminary stage, for high-risk groups, risky gaming behavior, gaming disorder layout hierarchical multidimensional assessment intervention system, using science education, brief intervention, social psychological intervention, neural regulation, cognitive rehabilitation training, mobile medical treatment, and other ways, stratification and stage, early identification, prevention and treatment combination, accurate intervention to comprehensively reduce the occurrence and development of gaming disorder.

ELIGIBILITY:
Inclusion Criteria:

* (1)Clinical diagnosis of severe Gaming Disorder defined in the ICD-11; (2)Normal hearing and vision, or within normal range after correction;

Exclusion Criteria:

* (1) Clinical diagnosis of mental health disorders other than GD defined in the ICD-11 in the past 5 years；(2) Suffering from diseases that affect cognitive function (such as cerebrovascular diseases) ; (3) Schizophrenia, bipolar disorder, depression or other Axis I disorder of DSM-V criteria;(4)any contraindication for tACS intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cue-induced craving | Two weeks,Four weeks
  Craving was assessed by visual analog scales (VAS), with 0 mm being "no craving"and 100 mm representing "most craving ever experienced for gaming ".
inter-brain synchronization (IBS) | Two weeks,Four weeks
  IBS was assessed by fNIRS hyperscanning with WTC analysis. A higher WTC refers to a higher level of inter-brain synchronization.
cognition measures | Four weeks
  Chinese version of the CogState Battery was used to assess cognitive function. We selected five tasks: Two back task (working memory), Continuous paired association task (visual spatial working memory), Groton maze learning task (error monitoring), social emotional cognition (social emotional cognition) and Detection task (processing speed) which were displayed on a green screen with standardized instructions before each task beginning.The accuracy in Two back task, social emotional cognition, and the speed in Detection task, and total errors in Continuous paired association task, Groton maze learning task are our focus.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China